CLINICAL TRIAL: NCT04685681
Title: Examining Adults' Activity Choices During COVID-19: The UB GO Study
Brief Title: The Get Outside Study
Acronym: GO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Stephanie Anzman-Frasca, Assistant Professor of Pediatrics, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005101
Record Dates: First submitted 2020-12-07; First posted 2020-12-28 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Covid19; Risk Reduction; Stress; Sleep
Keywords: Covid19; high-risk activities; low-risk activities; stress; sleep; adults
MeSH Terms: conditions — COVID-19; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hiking Challenge (Experimental): This group receives access to the local hiking challenge after completion of baseline measure
  Interventions: Behavioral: Hiking challenge
- Activity list (Active Comparator): This group receives access to a resource sheet with activity ideas after completion of baseline measure and does not receive the main resource of interest (hiking challenge) until after the post-test (delayed intervention)
  Interventions: Other: Activity list

INTERVENTIONS:
Behavioral: Hiking challenge — The main intervention of interest is the provision of free access to a local hiking challenge (which is provided following baseline assessments in the experimental group and after the conclusion of the study in the control group; $20 value). If participants choose to sign up for the free hiking challenge, they receive a list of local hikes/nature walks, accompanying maps, scavenger-hunt-like activities (finding a certain landmark on each hike), and the opportunity to earn prizes and engage with other hikers on social media.
  Arms: Hiking Challenge
Other: Activity list — The control group will receive a list of CDC-recommended activities following the baseline survey and will receive the hiking challenge as a delayed intervention following post-test.
  Arms: Activity list

SUMMARY:
The primary aim of this study is to examine whether lower-risk activities displace participation in higher-risk behaviors during COVID-19. Investigators will test this aim by promoting specific activities that are expected to be low-risk when it comes to COVID-19 transmission (e.g., participating in a hiking challenge) and assessing impacts on participants' activity choices. Investigators also aim to describe adults' activity participation during COVID-19 generally and to examine secondary outcomes, including reported stress and sleep.

DETAILED DESCRIPTION:
The primary aim of this study is to examine whether lower-risk activities displace participation in higher-risk behaviors during COVID-19. Investigators will test this aim by promoting specific activities that are expected to be low-risk when it comes to COVID-19 transmission and assessing impacts on participants' activity choices.

There will be two study groups, Group 1 and Group 2, each of which will complete 3 online surveys and will be provided with information on lower-risk activities to do during COVID-19. Random assignment to groups will occur after the completion of a baseline survey. Group 1 will receive free access to a local hiking challenge after completing their baseline survey and an information sheet with current CDC-recommended activities after post-test. Group 2 will receive the same resources, but in the opposite order. Therefore, surveys administered at midpoint (~6 weeks) and post-test (~12 weeks) will allow for a test of the effects of providing access to the hiking challenge on outcomes of interest.

If participants choose to sign up for the hiking challenge, they receive a list of local hikes/nature walks, accompanying maps, scavenger-hunt-like activities (finding a certain landmark on each hike), and the opportunity to earn prizes and engage with other hikers on social media. The primary outcome will be the activities in which participants engage. An adapted version of the Pleasant Activities list (Koks) will be used to assess activities participants have engaged in during the past 30 days at baseline, midpoint (~6 weeks), and post-test (~12 weeks). Current CDC guidance will be used to code activities as lower- and higher-risk anticipating the creation of an aggregate frequency of activities in each of the following categories: activities done outdoors alone or with members of the household (lower risk), activities done indoors alone or with members of the household (lower risk), activities done outdoors with others not in one's household (moderate risk), and activities done indoors with others not in one's household (higher risk). Adults' participation in different types of activities will also be summarized generally, in addition to specific activities of interest (e.g., the lower risk activities that are being targeted, like hiking; and activities that have received attention as being particularly higher risk, like indoor restaurant dining). Investigators will also examine impacts of the provision of the hiking challenge on secondary outcomes, including reported stress and sleep.

The study has the potential to shed light on displacement of higher-risk activities through promotion of lower-risk activities that could serve as substitutes. It also allows for an assessment of the impacts of the local hiking challenge on aspects of well-being. The first cohort of data collection for this study took place between January 2021-April 2021. A replication study was conducted in January 2022-April 2022. The details of the replication study were nearly identical, with one change being the provision of hiking equipment valued at ~$25 (microspikes for the Hiking Challenge intervention group and hiking socks for Activity List controls/the delayed intervention), a modification made based on barriers reported in the original study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English speaking
* Has online access
* Reports living in Western New York
* Interested in receiving "suggestions for ways to get outside, stay active, and stay busy" during COVID-19
* No health problems that preclude participation
* Not currently involved in regular (at least weekly) hikes/nature walks

Exclusion Criteria:

* Is under 18 years of age
* Not English speaking
* Does not have online access
* Does not report living in Western New York
* Is not interested in "suggestions for ways to get outside, stay active, and stay busy" during COVID-19
* Has health problems precluding participation
* Is currently involved in regular hikes/nature walks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Frequency of lower-risk activities | Post-test (12 weeks)
  Participants will indicate the frequency that they complete various activities using an adapted version of the Pleasant Activities List (Koks). Frequencies of each activity are indicated on a 0-4 scale where 0=never in the past 30 days and 4=very often in the past 30 days/more than 1 time per week. For each activity, participants will also indicate if it was done indoors or outdoors and who was there. We will aggregate the frequencies of activities that are lower-risk for COVID-19 transmission based on CDC recommendations at the time of the study. We anticipate that two indicators of lower-risk activities will be those completed outdoors by oneself or with individuals in the household and those completed indoors in which only the self or those in the household are present.
Frequency of higher-risk activities | Post-test (12 weeks)
  Participants will indicate the frequency that they complete various activities using an adapted version of the Pleasant Activities List (Koks). Frequencies of each activity are indicated on a 0-4 scale where 0=never in the past 30 days and 4=very often in the past 30 days/more than 1 time per week. For each activity, participants will also indicate if it was done indoors or outdoors and who was there. We will aggregate the frequencies of activities that are higher-risk for COVID-19 transmission based on CDC recommendations at the time of the study. We anticipate that two indicators of moderate- or high-risk activities will be those completed outdoors with individuals who do not live in one's household (moderate) and those completed indoors with individuals who do not live in one's household (high).
Frequency of social activities | Post-test (12 weeks)
  Participants will indicate the frequency that they complete various activities using an adapted version of the Pleasant Activities List (Koks). Frequencies of each activity are indicated on a 0-4 scale where 0=never in the past 30 days and 4=very often in the past 30 days/more than 1 time per week. For each activity, participants will also indicate if it was done indoors or outdoors and who was there. We will aggregate the frequencies of activities that are social, both those done with members of the household as well as those done with individuals who do not live in the household with the participant
Frequency of physical activities | Post-test (12 weeks)
  Participants will indicate the frequency that they complete various activities using an adapted version of the Pleasant Activities List (Koks). Frequencies of each activity are indicated on a 0-4 scale where 0=never in the past 30 days and 4=very often in the past 30 days/more than 1 time per week. For each activity, participants will also indicate if it was done indoors or outdoors and who was there. We will aggregate the frequencies of activities that involve physical activity (e.g., walks, hikes, sports)
Frequency of hiking/nature walks | Post-test (12 weeks)
  Participants will indicate the frequency that they complete various activities using an adapted version of the Pleasant Activities List (Koks). Frequencies of each activity are indicated on a 0-4 scale where 0=never in the past 30 days and 4=very often in the past 30 days/more than 1 time per week. For each activity, participants will also indicate if it was done indoors or outdoors and who was there. We will examine the frequency indicated for the item: Going on a hike or nature walk
Frequency of restaurant dining | Post-test (12 weeks)
  Participants will indicate the frequency that they complete various activities using an adapted version of the Pleasant Activities List (Koks). Frequencies of each activity are indicated on a 0-4 scale where 0=never in the past 30 days and 4=very often in the past 30 days/more than 1 time per week. For each activity, participants will also indicate if it was done indoors or outdoors and who was there. We will examine the frequency indicated for the item: Going to a restaurant or café / eating out

SECONDARY OUTCOMES:
Stress | Post-test (12 weeks)
  The 10-item perceived stress scale will be used to assess stress over the past month. Each item is scored from 0-4, for a total possible score of 0-40 (higher score = more stress).
Sleep | Post-test (12 weeks)
  Total nighttime sleep time will come from the Pittsburgh Sleep Quality Index (hours).

OTHER OUTCOMES:
Frequency of lower-risk activities | Midpoint (6 weeks)
  Participants will indicate the frequency that they complete various activities using an adapted version of the Pleasant Activities List (Koks). Frequencies of each activity are indicated on a 0-4 scale where 0=never in the past 30 days and 4=very often in the past 30 days/more than 1 time per week. For each activity, participants will also indicate if it was done indoors or outdoors and who was there. We will aggregate the frequencies of activities that are lower-risk for COVID-19 transmission based on CDC recommendations at the time of the study. We anticipate that two indicators of lower-risk activities will be those completed outdoors by oneself or with individuals in the household and those completed indoors in which only the self or those in the household are present.
Frequency of lower-risk activities | Change from baseline to post-test (12 weeks)
  Participants will indicate the frequency that they complete various activities using an adapted version of the Pleasant Activities List (Koks). Frequencies of each activity are indicated on a 0-4 scale where 0=never in the past 30 days and 4=very often in the past 30 days/more than 1 time per week. For each activity, participants will also indicate if it was done indoors or outdoors and who was there. We will aggregate the frequencies of activities that are lower-risk for COVID-19 transmission based on CDC recommendations at the time of the study. We anticipate that two indicators of lower-risk activities will be those completed outdoors by oneself or with individuals in the household and those completed indoors in which only the self or those in the household are present.
Frequency of higher-risk activities | Midpoint (6 weeks)
  Participants will indicate the frequency that they complete various activities using an adapted version of the Pleasant Activities List (Koks). Frequencies of each activity are indicated on a 0-4 scale where 0=never in the past 30 days and 4=very often in the past 30 days/more than 1 time per week. For each activity, participants will also indicate if it was done indoors or outdoors and who was there. We will aggregate the frequencies of activities that are higher-risk for COVID-19 transmission based on CDC recommendations at the time of the study. We anticipate that two indicators of moderate- or high-risk activities will be those completed outdoors with individuals who do not live in one's household (moderate) and those completed indoors with individuals who do not live in one's household (high).
Frequency of higher-risk activities | Change from baseline to post-test (12 weeks)
  Participants will indicate the frequency that they complete various activities using an adapted version of the Pleasant Activities List (Koks). Frequencies of each activity are indicated on a 0-4 scale where 0=never in the past 30 days and 4=very often in the past 30 days/more than 1 time per week. For each activity, participants will also indicate if it was done indoors or outdoors and who was there. We will aggregate the frequencies of activities that are higher-risk for COVID-19 transmission based on CDC recommendations at the time of the study. We anticipate that two indicators of moderate- or high-risk activities will be those completed outdoors with individuals who do not live in one's household (moderate) and those completed indoors with individuals who do not live in one's household (high).
Frequency of hiking/nature walks | Midpoint (6 weeks)
  Participants will indicate the frequency that they complete various activities using an adapted version of the Pleasant Activities List (Koks). Frequencies of each activity are indicated on a 0-4 scale where 0=never in the past 30 days and 4=very often in the past 30 days/more than 1 time per week. For each activity, participants will also indicate if it was done indoors or outdoors and who was there. Here we will examine responses to the item about the frequency of hiking or nature walks.
Frequency of hiking/nature walks | Change from baseline to post-test (12 weeks)
  Participants will indicate the frequency that they complete various activities using an adapted version of the Pleasant Activities List (Koks). Frequencies of each activity are indicated on a 0-4 scale where 0=never in the past 30 days and 4=very often in the past 30 days/more than 1 time per week. For each activity, participants will also indicate if it was done indoors or outdoors and who was there. Here we will examine responses to the item about the frequency of hiking or nature walks.
Stress | Midpoint (6 weeks)
  The 10-item perceived stress scale will be used to assess stress over the past month. Each item is scored from 0-4, for a total possible score of 0-40 (higher score = more stress).
Stress | Change from baseline to post-test (12 weeks)
  The 10-item perceived stress scale will be used to assess stress over the past month. Each item is scored from 0-4, for a total possible score of 0-40 (higher score = more stress).
Sleep | Midpoint (6 weeks)
  Total nighttime sleep time will come from the Pittsburgh Sleep Quality Index (hours).
Sleep | Change from baseline to post-test (12 weeks)
  Total nighttime sleep time will come from the Pittsburgh Sleep Quality Index (hours).

CONTACTS AND LOCATIONS:
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anzman-Frasca S, Drozdowsky J, Zayatz C, Holmbeck K. Effects of a randomized controlled hiking intervention on daily activities, sleep, and stress among adults during the COVID-19 pandemic. BMC Public Health. 2023 May 15;23(1):892. doi: 10.1186/s12889-023-15696-7. PMID 37189100